CLINICAL TRIAL: NCT07383454
Title: Lung Cancer Screening in Population Who Had Never Smoked and the Validation of Lung Cancer Risk Prediction Model
Brief Title: Lung Cancer Screening in Population Who Had Never Smoked
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Principal Investigator, Gee-Chen Chang, Professor, Chung Shan Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CS1-26008
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer (Diagnosis); Non-Small Cell Lung Cancer; Small Cell Carcinoma of Lung; Screening Strategy
Keywords: Low dose computed tomography (LDCT); Lung cancer in individuals who had never smoked (LCINS); Lung cancer risk prediction model (LCRPM); Lung cancer; Non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Disease; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDCT screening arm (Experimental): LDCT screening, lung function test, and specimens collections
  Interventions: Diagnostic Test: Low dose computed tomography

INTERVENTIONS:
Diagnostic Test: Low dose computed tomography — Low dose computed tomography for lung cancer screening

SUMMARY:
Study design: prospective, single arm.

Objectives: survey lung cancer detection rate of low-dose computed tomography (LDCT) screening in individuals who had never smoked.

Participants will undergo questionnaires, and collecting specimens including blood, urine, and medical informations including results of pulmonary function tests, and LDCT screening upon inclusion. The participants will be followed up according to current standards of clinical practice.

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-related mortality worldwide, with a particularly high incidence and mortality rate in Taiwan. Notably, over half of lung cancer cases in Taiwan occur among individuals who have never smoked, a pattern distinct from Western populations. In response to this unique epidemiological profile, this project aims to promote community-based lung cancer screening among never-smokers and to validate the FORMOSA lung cancer risk prediction model, which integrates demographic, environmental, genetic, and clinical factors.

This prospective, single-arm, open-label study will recruit approximately 2,500 participants aged 40 to 80 years with no history of smoking, through hospital and community outreach. Eligible participants will provide informed consent and undergo comprehensive assessments, including questionnaires on lifestyle and environmental exposures, low-dose computed tomography (LDCT), chest X-ray, pulmonary function tests, and collection of blood and urine samples. LDCT results will be interpreted according to the modified ACR Lung-RADS v1.1 criteria. Biological specimens will be used for biomarker, heavy metal, genetic, and proteomic analyses. Participants with abnormal findings will be followed according to standard clinical protocols, and tissue samples from invasive procedures will be retained for further molecular studies.

The primary outcomes include the lung cancer detection rate among never-smoked participants and the validation metrics (sensitivity, specificity, positive and negative predictive values) of the FORMOSA lung cancer risk prediction model. Statistical analyses will employ descriptive statistics, Kaplan-Meier survival analysis, log-rank tests, Cox proportional hazards models, and group comparisons using ANOVA, Kruskal-Wallis, chi-square, Fisher's exact tests, and logistic-regression. Preliminary data suggest that the FORMOSA model can identify high-risk individuals with a lung cancer detection rate of 2.8-3.3%, significantly higher than the general population rate of 0.78%.

This project is expected to enhance early detection of lung cancer in never-smokers, improve public awareness, and establish a robust epidemiological database for Taiwan. The validation of the FORMOSA model will provide a scientific basis for refining screening strategies and inform future public health policies targeting high-risk, non-smoking populations. The study is conducted with strict adherence to ethical standards, ensuring participant rights and data security. Funding is provided by the Ministry of Health and Welfare's "Healthy Taiwan Deep Cultivation Plan." In summary, this research addresses a critical gap in lung cancer prevention by focusing on never-smokers, leveraging a comprehensive risk prediction model, and implementing a community-based screening approach. The anticipated outcomes will contribute significantly to reducing late-stage lung cancer diagnoses and mortality, and serve as a reference for future health policy development in Taiwan and similar populations.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with no history of smoking.
2. Aged 40 to 80 years.
3. Willing to provide written informed consent and complete questionnaire assessments.
4. After undergoing examinations, willing to provide relevant biological information, including but not limited to: blood samples, urine samples, pulmonary function test results, imaging data, and tissue specimens obtained from invasive biopsies or surgical procedures (if applicable).

Exclusion Criteria:

1. History of lung cancer, or a diagnosis of any malignancy other than skin cancer or cervical carcinoma in situ within the past five years.
2. Undergoing chest computed tomography (CT) scans within the past 18 months.
3. Unexplained hemoptysis within the past one month.
4. Unexplained weight loss exceeding 6 kilograms within the past one year.
5. Pregnancy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Lung cancer detection rate | 8 years of follow-up
  The rate of lung cancer diagnosis during follow up periord.

SECONDARY OUTCOMES:
AUROC of FORMOSA Lung Cancer Risk Prediction Model | 8 years
  Assess the sensitivity, specificity, positive predicting value, negative predicting value, and ROC analysis of FORMOSA Lung Cancer Risk Prediction Model

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shi J, Shiraishi K, Choi J, Matsuo K, Chen TY, Dai J, Hung RJ, Chen K, Shu XO, Kim YT, Landi MT, Lin D, Zheng W, Yin Z, Zhou B, Song B, Wang J, Seow WJ, Song L, Chang IS, Hu W, Chien LH, Cai Q, Hong YC, Kim HN, Wu YL, Wong MP, Richardson BD, Funderburk KM, Li S, Zhang T, Breeze C, Wang Z, Blechter B, Bassig BA, Kim JH, Albanes D, Wong JYY, Shin MH, Chung LP, Yang Y, An SJ, Zheng H, Yatabe Y, Zhang XC, Kim YC, Caporaso NE, Chang J, Ho JCM, Kubo M, Daigo Y, Song M, Momozawa Y, Kamatani Y, Kobayashi M, Okubo K, Honda T, Hosgood DH, Kunitoh H, Patel H, Watanabe SI, Miyagi Y, Nakayama H, Matsumoto S, Horinouchi H, Tsuboi M, Hamamoto R, Goto K, Ohe Y, Takahashi A, Goto A, Minamiya Y, Hara M, Nishida Y, Takeuchi K, Wakai K, Matsuda K, Murakami Y, Shimizu K, Suzuki H, Saito M, Ohtaki Y, Tanaka K, Wu T, Wei F, Dai H, Machiela MJ, Su J, Kim YH, Oh IJ, Lee VHF, Chang GC, Tsai YH, Chen KY, Huang MS, Su WC, Chen YM, Seow A, Park JY, Kweon SS, Chen KC, Gao YT, Qian B, Wu C, Lu D, Liu J, Schwartz AG, Houlston R, Spitz MR, Gorlov IP, Wu X, Yang P, Lam S, Tardon A, Chen C, Bojesen SE, Johansson M, Risch A, Bickeboller H, Ji BT, Wichmann HE, Christiani DC, Rennert G, Arnold S, Brennan P, McKay J, Field JK, Shete SS, Le Marchand L, Liu G, Andrew A, Kiemeney LA, Zienolddiny-Narui S, Grankvist K, Johansson M, Cox A, Taylor F, Yuan JM, Lazarus P, Schabath MB, Aldrich MC, Jeon HS, Jiang SS, Sung JS, Chen CH, Hsiao CF, Jung YJ, Guo H, Hu Z, Burdett L, Yeager M, Hutchinson A, Hicks B, Liu J, Zhu B, Berndt SI, Wu W, Wang J, Li Y, Choi JE, Park KH, Sung SW, Liu L, Kang CH, Wang WC, Xu J, Guan P, Tan W, Yu CJ, Yang G, Sihoe ADL, Chen Y, Choi YY, Kim JS, Yoon HI, Park IK, Xu P, He Q, Wang CL, Hung HH, Vermeulen RCH, Cheng I, Wu J, Lim WY, Tsai FY, Chan JKC, Li J, Chen H, Lin HC, Jin L, Liu J, Sawada N, Yamaji T, Wyatt K, Li SA, Ma H, Zhu M, Wang Z, Cheng S, Li X, Ren Y, Chao A, Iwasaki M, Zhu J, Jiang G, Fei K, Wu G, Chen CY, Chen CJ, Yang PC, Yu J, Stevens VL, Fraumeni JF Jr, Chatterjee N, Gorlova OY, Hsiung CA, Amos CI, Shen H, Chanock SJ, Rothman N, Kohno T, Lan Q. Genome-wide association study of lung adenocarcinoma in East Asia and comparison with a European population. Nat Commun. 2023 May 26;14(1):3043. doi: 10.1038/s41467-023-38196-z. PMID 37236969
- [Background] Diaz-Gay M, Zhang T, Hoang PH, Leduc C, Baine MK, Travis WD, Sholl LM, Joubert P, Khandekar A, Zhao W, Steele CD, Otlu B, Nandi SP, Vangara R, Bergstrom EN, Kazachkova M, Pich O, Swanton C, Hsiung CA, Chang IS, Wong MP, Leung KC, Sang J, McElderry JP, Hartman C, Colon-Matos FJ, Miraftab M, Saha M, Lee OW, Jones KM, Gallego-Garcia P, Yang Y, Zhong X, Edell ES, Santamaria JM, Schabath MB, Yendamuri SS, Manczuk M, Lissowska J, Swiatkowska B, Mukeria A, Shangina O, Zaridze D, Holcatova I, Mates D, Milosavljevic S, Kontic M, Bosse Y, Rothberg BEG, Christiani DC, Gaborieau V, Brennan P, Liu G, Hofman P, Yang L, Nowak MA, Shi J, Rothman N, Wedge DC, Homer R, Yang SR, Pesatori AC, Consonni D, Lan Q, Zhu B, Chanock SJ, Choi J, Alexandrov LB, Landi MT. The mutagenic forces shaping the genomes of lung cancer in never smokers. Nature. 2025 Aug;644(8075):133-144. doi: 10.1038/s41586-025-09219-0. Epub 2025 Jul 2. PMID 40604281
- [Background] Chen IC, Chen YM, Yang HW, Tseng JS, Yang TY. Interplay of Polygenic Risk Score, Smoking Statuses, and Air Pollution on Lung Adenocarcinoma Risk in a Taiwanese Population. Respirology. 2025 Apr;30(4):317-325. doi: 10.1111/resp.70004. Epub 2025 Feb 16. PMID 39956994
- [Background] Blechter B, Chien LH, Chen TY, Chang IS, Choudhury PP, Hsiao CF, Shu XO, Wong JYY, Chen KY, Chang GC, Tsai YH, Su WC, Huang MS, Chen YM, Chen CY, Hung HH, Hu JW, Shi J, Zheng W, Rositch AF, Chen CJ, Chatterjee N, Yang PC, Rothman N, Hsiung CA, Lan Q. Polygenic Risk Score, Environmental Tobacco Smoke, and Risk of Lung Adenocarcinoma in Never-Smoking Women in Taiwan. JAMA Netw Open. 2023 Nov 1;6(11):e2339254. doi: 10.1001/jamanetworkopen.2023.39254. PMID 37955902
- [Background] Blechter B, Wong JYY, Agnes Hsiung C, Hosgood HD, Yin Z, Shu XO, Zhang H, Shi J, Song L, Song M, Zheng W, Wang Z, Caporaso N, Burdette L, Yeager M, Berndt SI, Teresa Landi M, Chen CJ, Chang GC, Hsiao CF, Tsai YH, Chen KY, Huang MS, Su WC, Chen YM, Chien LH, Chen CH, Yang TY, Wang CL, Hung JY, Lin CC, Perng RP, Chen CY, Chen KC, Li YJ, Yu CJ, Chen YS, Chen YH, Tsai FY, Jie Seow W, Bassig BA, Hu W, Ji BT, Wu W, Guan P, He Q, Gao YT, Cai Q, Chow WH, Xiang YB, Lin D, Wu C, Wu YL, Shin MH, Hong YC, Matsuo K, Chen K, Pik Wong M, Lu D, Jin L, Wang JC, Seow A, Wu T, Shen H, Fraumeni JF, Yang PC, Chang IS, Zhou B, Chanock SJ, Rothman N, Chatterjee N, Lan Q. Sub-multiplicative interaction between polygenic risk score and household coal use in relation to lung adenocarcinoma among never-smoking women in Asia. Environ Int. 2021 Feb;147:105975. doi: 10.1016/j.envint.2020.105975. Epub 2020 Dec 29. PMID 33385923
- [Background] Coradduzza D, Congiargiu A, Azara E, Mammani IMA, De Miglio MR, Zinellu A, Carru C, Medici S. Heavy metals in biological samples of cancer patients: a systematic literature review. Biometals. 2024 Aug;37(4):803-817. doi: 10.1007/s10534-024-00583-4. Epub 2024 Feb 12. PMID 38347295
- [Background] Lee NW, Wang HY, Du CL, Yuan TH, Chen CY, Yu CJ, Chan CC. Air-polluted environmental heavy metal exposure increase lung cancer incidence and mortality: A population-based longitudinal cohort study. Sci Total Environ. 2022 Mar 1;810:152186. doi: 10.1016/j.scitotenv.2021.152186. Epub 2021 Dec 6. PMID 34883183
- [Background] Huang HH, Huang JY, Lung CC, Wu CL, Ho CC, Sun YH, Ko PC, Su SY, Chen SC, Liaw YP. Cell-type specificity of lung cancer associated with low-dose soil heavy metal contamination in Taiwan: an ecological study. BMC Public Health. 2013 Apr 10;13:330. doi: 10.1186/1471-2458-13-330. PMID 23575356
- [Background] Yoon HY, Kim SY, Song JW. Association between high levels of nitrogen dioxide and increased cumulative incidence of lung cancer in patients with idiopathic pulmonary fibrosis. Eur Respir J. 2024 May 30;63(5):2301181. doi: 10.1183/13993003.01181-2023. Print 2024 May. PMID 38453259
- [Background] Hamra GB, Laden F, Cohen AJ, Raaschou-Nielsen O, Brauer M, Loomis D. Lung Cancer and Exposure to Nitrogen Dioxide and Traffic: A Systematic Review and Meta-Analysis. Environ Health Perspect. 2015 Nov;123(11):1107-12. doi: 10.1289/ehp.1408882. Epub 2015 Apr 14. PMID 25870974
- [Background] Lin WC, Shie RH, Yuan TH, Tseng CH, Chiang CJ, Lee WC, Chan CC. A nationwide case-referent study on elevated risks of adenocarcinoma lung cancer by long-term PM2.5 exposure in Taiwan since 1997. Environ Res. 2024 Jul 1;252(Pt 2):118889. doi: 10.1016/j.envres.2024.118889. Epub 2024 Apr 8. PMID 38599452
- [Background] Jones RR, Fisher JA, Hasheminassab S, Kaufman JD, Freedman ND, Ward MH, Sioutas C, Vermeulen R, Hoek G, Silverman DT. Outdoor Ultrafine Particulate Matter and Risk of Lung Cancer in Southern California. Am J Respir Crit Care Med. 2024 Feb 1;209(3):307-315. doi: 10.1164/rccm.202305-0902OC. PMID 37856832
- [Background] Hill W, Lim EL, Weeden CE, Lee C, Augustine M, Chen K, Kuan FC, Marongiu F, Evans EJ Jr, Moore DA, Rodrigues FS, Pich O, Bakker B, Cha H, Myers R, van Maldegem F, Boumelha J, Veeriah S, Rowan A, Naceur-Lombardelli C, Karasaki T, Sivakumar M, De S, Caswell DR, Nagano A, Black JRM, Martinez-Ruiz C, Ryu MH, Huff RD, Li S, Fave MJ, Magness A, Suarez-Bonnet A, Priestnall SL, Luchtenborg M, Lavelle K, Pethick J, Hardy S, McRonald FE, Lin MH, Troccoli CI, Ghosh M, Miller YE, Merrick DT, Keith RL, Al Bakir M, Bailey C, Hill MS, Saal LH, Chen Y, George AM, Abbosh C, Kanu N, Lee SH, McGranahan N, Berg CD, Sasieni P, Houlston R, Turnbull C, Lam S, Awadalla P, Gronroos E, Downward J, Jacks T, Carlsten C, Malanchi I, Hackshaw A, Litchfield K; TRACERx Consortium; DeGregori J, Jamal-Hanjani M, Swanton C. Lung adenocarcinoma promotion by air pollutants. Nature. 2023 Apr;616(7955):159-167. doi: 10.1038/s41586-023-05874-3. Epub 2023 Apr 5. PMID 37020004
- [Background] Loomis D, Huang W, Chen G. The International Agency for Research on Cancer (IARC) evaluation of the carcinogenicity of outdoor air pollution: focus on China. Chin J Cancer. 2014 Apr;33(4):189-96. doi: 10.5732/cjc.014.10028. PMID 24694836
- [Background] Loomis D, Grosse Y, Lauby-Secretan B, El Ghissassi F, Bouvard V, Benbrahim-Tallaa L, Guha N, Baan R, Mattock H, Straif K; International Agency for Research on Cancer Monograph Working Group IARC. The carcinogenicity of outdoor air pollution. Lancet Oncol. 2013 Dec;14(13):1262-3. doi: 10.1016/s1470-2045(13)70487-x. No abstract available. PMID 25035875
- [Background] Wang CL, Hsu KH, Chang YH, Ho CC, Chiang CJ, Chen KC, Cheung YC, Huang PC, Chen YR, Chen CY, Hsu CP, Hsia JY, Chen HY, Yang SY, Li YJ, Yang TY, Tseng JS, Chuang CY, Hsiung CA, Chen YM, Huang MS, Yu CJ, Chen KY, Su WC, Chen JJW, Yu SL, Chen CJ, Yang PC, Tsai YH, Chang GC. Low-Dose Computed Tomography Screening in Relatives With a Family History of Lung Cancer. J Thorac Oncol. 2023 Nov;18(11):1492-1503. doi: 10.1016/j.jtho.2023.06.018. Epub 2023 Jul 5. PMID 37414358
- [Background] Lo YL, Hsiao CF, Chang GC, Tsai YH, Huang MS, Su WC, Chen YM, Hsin CW, Chang CH, Yang PC, Chen CJ, Hsiung CA. Risk factors for primary lung cancer among never smokers by gender in a matched case-control study. Cancer Causes Control. 2013 Mar;24(3):567-76. doi: 10.1007/s10552-012-9994-x. Epub 2012 May 22. PMID 22729933
- [Background] Murphy C, Pandya T, Swanton C, Solomon BJ. Lung Cancer in Nonsmoking Individuals: A Review. JAMA. 2025 Nov 25;334(20):1836-1845. doi: 10.1001/jama.2025.17695. PMID 41114991
- [Background] Chang GC, Chiu CH, Yu CJ, Chang YC, Chang YH, Hsu KH, Wu YC, Chen CY, Hsu HH, Wu MT, Yang CT, Chong IW, Lin YC, Hsia TC, Lin MC, Su WC, Lin CB, Lee KY, Wei YF, Lan GY, Chan WP, Wang KL, Wu MH, Tsai HH, Chian CF, Lai RS, Shih JY, Wang CL, Hsu JS, Chen KC, Chen CK, Hsia JY, Peng CK, Tang EK, Hsu CL, Chou TY, Shen WC, Tsai YH, Tsai CM, Chen YM, Lee YC, Chen HY, Yu SL, Chen CJ, Wan YL, Hsiung CA, Yang PC; TALENT Investigators. Low-dose CT screening among never-smokers with or without a family history of lung cancer in Taiwan: a prospective cohort study. Lancet Respir Med. 2024 Feb;12(2):141-152. doi: 10.1016/S2213-2600(23)00338-7. Epub 2023 Nov 29. PMID 38042167
- [Background] Tseng CH, Tsuang BJ, Chiang CJ, Ku KC, Tseng JS, Yang TY, Hsu KH, Chen KC, Yu SL, Lee WC, Liu TW, Chan CC, Chang GC. The Relationship Between Air Pollution and Lung Cancer in Nonsmokers in Taiwan. J Thorac Oncol. 2019 May;14(5):784-792. doi: 10.1016/j.jtho.2018.12.033. Epub 2019 Jan 18. PMID 30664991
- [Background] Lam DC, Liam CK, Andarini S, Park S, Tan DSW, Singh N, Jang SH, Vardhanabhuti V, Ramos AB, Nakayama T, Nhung NV, Ashizawa K, Chang YC, Tscheikuna J, Van CC, Chan WY, Lai YH, Yang PC. Lung Cancer Screening in Asia: An Expert Consensus Report. J Thorac Oncol. 2023 Oct;18(10):1303-1322. doi: 10.1016/j.jtho.2023.06.014. Epub 2023 Jun 28. PMID 37390982
- [Background] Wolf AMD, Oeffinger KC, Shih TY, Walter LC, Church TR, Fontham ETH, Elkin EB, Etzioni RD, Guerra CE, Perkins RB, Kondo KK, Kratzer TB, Manassaram-Baptiste D, Dahut WL, Smith RA. Screening for lung cancer: 2023 guideline update from the American Cancer Society. CA Cancer J Clin. 2024 Jan-Feb;74(1):50-81. doi: 10.3322/caac.21811. Epub 2023 Nov 1. PMID 37909877
- See also: Related Info — https://www.airitilibrary.com/Article/Detail?DocID=17263603-N202505200008-00005